CLINICAL TRIAL: NCT02986308
Title: The Metabolomics of Intestinal Polyps of Different Pathological Types and TCM Syndromes and TCM Constitution Types
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wei Xu, MD,Professor, First Affiliated Hospital of Harbin Medical University
Other Study IDs: Wei Xu
Record Dates: First submitted 2016-08-01; First posted 2016-12-08 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Intestinal Polyps
Keywords: Metabolomics; Intestinal Polyps; TCM Syndromes; TCM Constitution Types
MeSH Terms: conditions — Intestinal Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples With DNA — serum

GROUPS / COHORTS (2):
- Intestinal Polyps: The patients who were diagnosed with Intestinal Polyps.
  Interventions: Other: No intervention
- Normal colonoscopy: People who were diagnosed by colonoscopy without intestinal polyps.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The aim of this study is to confirm the TCM syndrome types and TCM constitution classifications of the patients with intestinal polyps via on-site epidemiological survey, to analyze metabolomics of the serum samples of intestinal polyps and healthy volunteers, and to study the metabolomics differences of the two populations and the metabolomics variations of the patients with intestinal polyps of pre-polypectomy and post-polypectomy. Finally, this study is to investigate the serum metabolomics variations of patients with intestinal polyps of pre-polypectomy and post-polypectomy and the relationship with their TCM syndrome types and TCM constitution classifications, to determine the correlation among pathology, TCM constitution, TCM syndrome types and the metabonomics variations of patients with intestinal polyps.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 to 80,all genders;
2. Intestinal polyps were found by colonoscopy;
3. The patients are scheduled for polypectomy;
4. Preoperative examinations were completed;
5. Performance status 0-1;
6. Diet has well controlled prior to the operation;
7. Patients or their statutory agent have signed the informed consent forms.

Exclusion Criteria:

1. The patient has not diagnosed by colonoscopy;
2. The patient has surgical contraindication;
3. Patients in pregnant or lactational period ;
4. Psychopath;
5. The patient is in drug trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intestinal polyps patients
Sampling Method: Non-Probability Sample
Enrollment: 1659 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Aiming to obtain biomarker groups of different pathological types of intestinal polyps, The potential biomarkers will be entered KEGG database to obtain metabolic pathways. | 2 years

SECONDARY OUTCOMES:
All data matrices are introduced to Ezinfo software for PCA and OPLS-DA. Using improved "MetPA enriched pathways" method to discover the metabolic pathways of the disease. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Doctor, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Du WZ, Zhang AH, Ren JL, Lyu K, Tuo LY, Xu W. Study of Differential Serum Metabolites in Patients with Adenomatous Polyps of Colon and Yang-Deficiency Constitution Based on Ultra-Performance Liquid Chromatography-Mass Spectrometry. Chin J Integr Med. 2022 May;28(5):403-409. doi: 10.1007/s11655-019-3181-9. Epub 2019 Nov 29. PMID 31784934